CLINICAL TRIAL: NCT07252804
Title: Short- and Long-Term Immunogenicity and Safety of Meningococcal Group B Vaccine in Children and Adolescents With Autoimmune Rheumatic Diseases
Brief Title: Immunogenicity and Safety of MenB Vaccine in Pediatric Patients With Autoimmune Rheumatic Diseases
Acronym: MENB-PARD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Insituto Adolfo Lutz (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 761245237 0000 0068
Record Dates: First submitted 2025-07-18; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Autoimmune Rheumatologic Disease
Keywords: Meningococcal B vaccine; Autoimmune Rheumatic Diseases; Rheumatology; Pediatric Rheumatology; Infectious Disease Prevention
MeSH Terms: interventions — 4CMenB vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- J-ARDs (Experimental): Patients with ARDs will receive 2 doses (0.5 mL each) of Bexsero, 1 month apart
  Interventions: Biological: Meningococcal B (Bexsero)
- Control (Active Comparator): Healthy participants will receive 2 doses (0.5 mL each) of Bexsero, 1 month apart
  Interventions: Biological: Meningococcal B (Bexsero)

INTERVENTIONS:
Biological: Meningococcal B (Bexsero) — The MenB-4C vaccine consists of three recombinant antigenic proteins: Neisseria meningitidis Neisseria adhesin A (NadA), factor H binding protein subfamily B (FHbp-B), and Neisseria heparin-binding antigen (NHBA), along with outer membrane vesicles (OMVs) expressing porin A (PorA) protein from serosubtype P1.4. The MenB-4C vaccine will be administered intramuscularly (into the deltoid muscle) in 2 doses of 0.5 mL each, one month apart.
  Other Names: MenB-4C

SUMMARY:
The goal of this clinical trial is to evaluate the humoral immunogenicity of the meningococcal B vaccine (MenB-4C) in pediatric patients with autoimmune rheumatic diseases (ARDs), compared to age- and sex-matched non-immunosuppressed controls.

The main questions it aims to answer are:

* To assess the influence of treatment on the response to the MenB-4C vaccine in patients with ARDs;
* To evaluate the impact of the MenB-4C vaccine on disease activity in patients with ARDs;
* To evaluate the safety of the MenB-4C vaccine in pediatric patients with ARDs and controls.
* To evaluate the association between physical activity levels and immunogenicity after vaccination.

Participants will:

Receive the MenB-4C vaccine (Bexsero©), administered intramuscularly in the deltoid muscle, in a 2-dose schedule (0.5 mL each), 1 month apart.

All participants will have blood samples collected immediately before vaccination at the baseline visit (D0), then receive the first vaccine dose on the same day (D0). The second dose will be administered 4 weeks after the first dose (D28). Blood samples will be collected on D0, D28, and D56. A final sample will be collected one year after the last dose (D208) to evaluate the persistence of immune response.

At study entry and one month after each dose, patients will also be assessed for clinical and laboratory disease activity using disease-specific indices and scores.

* Juvenile Systemic lupus erythematosus (JSLE): Systemic lupus erythematosus disease activity index 2000 (SLEDAI-2K) (CBC, anti-dsDNA, complement, urinalysis, protein/creatinine ratio)
* Juvenile Idiopatic Arthritis (JIA): Juvenile Arthritis Disease Activity Score (JADAS) (ESR, CRP)
* Juvenile dermatomyositis (JDM): Manual Muscle Testing (MMT) e Childhood Myositis Assessment Scale (CMAS): (CPK, transaminases, LDH)

Researcher will also perform analysis in:

Humoral immunogenicity will be assessed using serum bactericidal activity (SBA) assay with exogenous complement (baby rabbit, Pel Freez) against four test strains: H44/76 (fHBP), 5/99 (NadA), NZ98/254 (PorA), and M10713 (NHBA), from blood samples collected at D0, D28, D56, and D208. SBA assays will be conducted at the Immunology Center of the Adolfo Lutz Institute, São Paulo. Exogenous complement will be added to serially diluted serum samples, followed by the addition of a bacterial suspension. The humoral response rate induced by the vaccine, or seroconversion, will be defined by the bactericidal titer (the dilution that results in 50% bacterial killing within 60 minutes compared to the control), with titers ≥ 1:4 considered bactericidal. The geometric mean titers will be calculated using the exponential of the mean of the log-transformed concentrations.

Immunosuppressive treatments (NSAIDs, prednisone/prednisolone, intra-articular steroids, hydroxychloroquine, methotrexate, azathioprine, leflunomide, cyclosporine, tacrolimus, mycophenolate mofetil, and biologics [anti-TNF, tocilizumab, abatacept, belimumab, rituximab]) will be recorded sistematicaly.

Physical activity levels will be assessed using validated, age-appropriate methods.

DETAILED DESCRIPTION:
Invasive meningococcal disease (IMD) is a severe infection caused by Neisseria meningitidis and can be life-threatening. In Brazil, the incidence of IMD has been reported as 2 per 100,000 children and adolescents, with serogroups B and C being the most prevalent. Severe infections are a major concern in patients with autoimmune rheumatic diseases (ARDs), as they are recognized as a leading cause of morbidity and mortality, accounting for up to one-third of all deaths in this population.

In this context, there are currently two licensed vaccines against serogroup B in Brazil: the MenB-4C vaccine (Bexsero©) by GlaxoSmithKline (GSK), which includes four components, and the MenB-FHbp vaccine (Trumenba©) by Pfizer, which includes two components. The MenB-4C (Bexsero©) vaccine has broader coverage and is recommended in Brazil from 2 months of age. MenB-FHbp (Trumenba©, Pfizer) is approved in Brazil only for adolescents and young adults aged 10 to 25 years. Neither of these vaccines is included in Brazil's National Immunization Program (PNI) due to their high cost.

Currently, the MenB-4C vaccine is licensed in over 35 countries and consists of three recombinant antigenic proteins. The Brazilian Society of Pediatrics recommends MenB-4C vaccination for children and adolescents aged 2 to 18 years, administered in two doses at least one month apart.

The immunogenicity and safety of MenB-4C has been demonstrated in the general population through a meta-analysis of 18 studies, including phase I, II, and III randomized controlled clinical trials, involving 6,637 children and adolescents aged 2 months to 17 years. The incidence of serious adverse events (SAEs) potentially related to the vaccine was very low (0.54%) but significantly higher than in controls (0.12%) who received routine childhood vaccines. Despite this, the safety profile of MenB-4C is considered acceptable.

Physical activity is a low-cost, scalable behavioral intervention that may enhance immune function, particularly relevant in immunocompromised populations such as children and adolescents with ARDs. While higher physical activity levels have been linked to improved vaccine responses in adults, its role in pediatric ARD patients remains unexplored. This study aims to fill this knowledge gap by investigating the association between physical activity and the humoral immune response to the MenB-4C vaccine, using both subjective and objective assessment methods.

However, to date, no studies have evaluated the immunogenicity, safety and physical activity levels after MenB vaccines in pediatric patients with ARDs.

Our study is a prospective, controlled, phase IV study that aims to evaluate the humoral immunogenicity of the MenB-4C vaccine in pediatric patients with ARDs compared to age and sex matched non-immunosuppressed controls. As secondary objectives we will assess the influence of short- and long-term immunosuppressive treatment on the vaccine response in patients with ARDs; to evaluate the impact of vaccination on disease activity in patients with ARDs; to assess the safety of the vaccine in pediatric ARD patients and controls and to evaluate the association between physical activity levels and vaccine-induced humoral immune responses in patients with ARDs.

Participants will be between 2 and 25 years of age. Patients with JIA will be diagnosed based on the classification criteria of the International League of Associations for Rheumatology (ILAR); patients with JSLE, according to the American College of Rheumatology (ACR); and those with JDM, according to Bohan & Peter criteria. A total of 263 patients will be included, of these,197 with ARDs and 66 healthy-matched controls.

All participants will receive the MenB-4C vaccine (Bexsero©), administered intramuscularly in the deltoid muscle, in two doses (0.5 mL each) one month apart.

Blood samples will be collected immediately before vaccination at baseline (D0), and the first vaccine dose will be administered on the same day (D0). The second dose will be administered 4 weeks after the first dose (D28). Blood samples will be collected on D0, D28, and D56. A final sample will be collected one year after the last dose (D208) to assess the persistence of the immune response.

At baseline and one month after each dose, patients will also be assessed for clinical and laboratory disease activity using disease-specific inflammatory activity indices:

* JSLE: Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K): complete blood count (hemoglobin in g/dL, white blood cells and platelets in 1000/mm3, anti-dsDNA antibodies (in UI/mL), complement (in mg/dL), urinalysis (heme-granular or red blood cells urinary casts, hematuria >5RBC/higpower field, proteinuria >0.5g/24 hours, pyuria (>5 white blood cells/ high-power field) and urine protein/creatinine ratio (in mg/dL);
* JIA: Juvenile Arthritis Disease Activity Score (JADAS): erythrocyte sedimentation rate (in mm), and C-reactive protein (in mg/L);
* JDM: Manual Muscle Testing (MMT) and Childhood Myositis Assessment Scale (CMAS): creatine phosphokinase (in U/L), transaminases (in U/L), and lactate dehydrogenase (in U/L).

Safety will be closely monitored, and all serious adverse events will be classified as related or unrelated to the vaccine. A standardized adverse event diary will be provided to all patients and healthy controls for recording local and systemic reactions during the 4 weeks following each vaccine dose (D28 and D56). Local reactions include: injection site pain, redness, swelling, bruising, itching, and induration. Systemic reactions include: fever, fatigue, chills, malaise, drowsiness, loss of appetite, nausea, vomiting, diarrhea, abdominal pain, dizziness, tremors, headache, fatigue, myalgia, muscle weakness, arthralgia, pruritus, and skin rash.

The severity of adverse events will be determined according to World Health Organization (WHO) criteria.

Immunosuppressive treatments at each time point-including nonsteroidal anti-inflammatory drugs, prednisone/prednisolone, intra-articular corticosteroids, hydroxychloroquine, methotrexate, azathioprine, leflunomide, cyclosporine, tacrolimus, mycophenolate mofetil, and biologics (anti-TNF, tocilizumab, abatacept, belimumab, and rituximab) -will be systematically evaluated and correlated with possible impact with seroconversion.

Humoral immunogenicity will be assessed by serum bactericidal activity (SBA) assay using exogenous complement (Baby rabbit, Pel Freez) against four test strains: H44/76 (fHBP), 5/99 (NadA), NZ98/254 (PorA), and M10713 (NHBA), from blood samples collected at D0, D30, D60, and D208. SBA assays will be performed at the Immunology Center of the Adolfo Lutz Institute, São Paulo.

Briefly, exogenous complement will be added to serially diluted serum samples, followed by the addition of a bacterial suspension. The humoral response rate induced by the vaccine, or seroconversion, will be defined by the bactericidal titer (the dilution that results in 50% bacterial killing within 60 minutes compared to the control), with titers ≥ 1:4 considered bactericidal. The geometric mean titers will be calculated using the exponential of the mean of the log-transformed concentrations.

Physical activity will be evaluated using age-appropriate validated questionnaires (IPAQ, PAQ-A, PAQ-C), classifying participants as active or inactive based on WHO guidelines (≥150 minutes/week of moderate-to-vigorous activity). Additionally, participants will wear a triaxial accelerometer (ActiGraph GTex®) continuously between days 7 and 14 after the first vaccine dose to objectively record movement intensity and volume.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between 2 and 25 years of age with no prior history of MenB-4C vaccination.
* Patients classified with autoimmune rheumatic diseases will be invited to participate.

Patients with JIA must meet the classification criteria of the International League of Associations for Rheumatology; patients with JSLE, the American College of Rheumatology criteria; and those with JDM, the Bohan & Peter criteria.

Exclusion Criteria:

* History of any reaction or hypersensitivity to any vaccine component;
* Acute infectious disease and/or fever at the time of vaccination;
* Pregnancy or breastfeeding;
* History of Guillain-Barré syndrome;
* Participants who fail to attend evaluation visits and laboratory sample collection; hospitalization at study inclusion;
* Transfusion of blood products within 6 months prior to the study;
* Application of any vaccine within one month prior to each dose.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 263 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Seroconversion Rate After Vaccination | Day 28 to Day 208
  Proportion of participants who achieve seroconversion. The humoral response rate induced by the vaccine, or seroconversion, will be defined by the bactericidal titer (the dilution resulting in 50% bacterial killing within 60 minutes compared to the control). Titers ≥ 1:4 will be considered bactericidal. The geometric mean titer will be calculated using the exponential of the mean of log-transformed concentrations.

SECONDARY OUTCOMES:
Influence of Immunosuppressive Treatment on the response to MenB-4C vaccination | Day 28 to Day 208
  To assess the short- and long-term influence of immunosuppressive treatment on the response to MenB-4C vaccination in patients with ARDs compared to healthy controls. Humoral immunogenicity will be evaluated using the serum bactericidal activity (SBA) assay with exogenous complement (Baby rabbit, Pel Freez) against 4 test strains: H44/76 (fHBP vaccine antigen evaluation), 5/99 (Neisseria adhesin A), NZ98/254 (Porin A) and M10713 (NHBA).
Impact of MenB-4C vaccination on Disease Activity on patients with JIA | Day 1 through D56
  To evaluate the impact of MenB-4C vaccination on clinical disease activity in patients with JIA, measured using JADAS27, higher scores indicates greater disease activity.
  Unit of Measure: Score (0-57).
Impact of MenB-4C vaccination on Disease Activity on patients with JSLE | Day 1 through Day 56
  To evaluate the impact of MenB-4C vaccination on clinical and laboratory disease activity in patients with juvenile systemic lupus erythematosus (jSLE), assessed using the SLEDAI-2K. The score incorporates clinical and laboratory manifestations of lupus, with higher scores indicating greater disease activity.
  Unit of Measure: Score (range 0-105).
Impact of MenB-4c vaccination on Disease Activity on patients with JDM | Day 1 through Day 56
  To evaluate the impact of MenB-4C vaccination on clinical and laboratory disease activity in patients with juvenile dermatomyositis (JDM), assessed using the Childhood Myositis Assessment Scale (CMAS). The CMAS evaluates muscle function and endurance, with higher scores indicating better muscle strength and physical performance.
  Unit of Measure: Score (range 0-52).
Number of patients with adverse events related to the vaccination with MenB-4C | Day 1 through Day 56
  Safety will be closely monitored, and all serious adverse events will be classified as related or unrelated to the vaccine. A standardized adverse event diary will be provided to all patients and healthy controls for recording local and systemic reactions during the 4 weeks following each vaccine dose. Local reactions include: injection site pain, redness, swelling, bruising, itching, and induration. Systemic reactions include: fever, fatigue, chills, malaise, drowsiness, loss of appetite, nausea, vomiting, diarrhea, abdominal pain, dizziness, tremors, headache, fatigue, myalgia, muscle weakness, arthralgia, pruritus, and skin rash.
Seroconversion Rates after MenB-4C vaccination by Physical Activity Classification | Day 1 to 208 post-vaccination
  Proportion of participants who achieve higher seroconversion rates and bactericidal titers (SBA) against vaccine-targeted strains concentrations compared to baseline at Days 28 and 180 following vaccination. Participants will be categorized as physically active or inactive based on World Health Organization criteria using validated methods.
Geometric mean titers of human serum bactericidal antibodies after the MenB-4C Vaccination by Physical Activity Classification | Day 1 to 208 post-vaccination
  Geometric mean titers of human serum bactericidal antibodies against the four reference MenB strains (H44/76, 5/99, NZ98/254, and M10713) will be measured at Days 28, 56, and 208 following MenB-4C vaccination. Participants will be classified as physically active or inactive based on World Health Organization criteria, based on validated methods.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perez-Vilar S, Dores GM, Marquez PL, Ng CS, Cano MV, Rastogi A, Lee L, Su JR, Duffy J. Safety surveillance of meningococcal group B vaccine (Bexsero(R)), Vaccine Adverse Event Reporting System, 2015-2018. Vaccine. 2022 Jan 21;40(2):247-254. doi: 10.1016/j.vaccine.2021.11.071. Epub 2021 Dec 7. PMID 34887130
- [Background] Flacco ME, Manzoli L, Rosso A, Marzuillo C, Bergamini M, Stefanati A, Cultrera R, Villari P, Ricciardi W, Ioannidis JPA, Contopoulos-Ioannidis DG. Immunogenicity and safety of the multicomponent meningococcal B vaccine (4CMenB) in children and adolescents: a systematic review and meta-analysis. Lancet Infect Dis. 2018 Apr;18(4):461-472. doi: 10.1016/S1473-3099(18)30048-3. Epub 2018 Jan 19. PMID 29371070
- [Background] Singh JA, Cleveland JD. Hospitalized Infections in Lupus: A Nationwide Study of Types of Infections, Time Trends, Health Care Utilization, and In-Hospital Mortality. Arthritis Rheumatol. 2021 Apr;73(4):617-630. doi: 10.1002/art.41577. Epub 2021 Mar 5. PMID 33142044
- [Background] Safadi MA, O'Ryan M, Valenzuela Bravo MT, Brandileone MC, Gorla MC, de Lemos AP, Moreno G, Vazquez JA, Lopez EL, Taha MK, Borrow R; Global Meningococcal Initiative. The current situation of meningococcal disease in Latin America and updated Global Meningococcal Initiative (GMI) recommendations. Vaccine. 2015 Nov 27;33(48):6529-36. doi: 10.1016/j.vaccine.2015.10.055. Epub 2015 Oct 25. PMID 26597036